CLINICAL TRIAL: NCT04212494
Title: Thrombus Aspiration in Primary Percutaneous Coronary Intervention for STEMI Patients With High Thrombus Burden
Brief Title: Thrombus Aspiration in STEMI Patients With High Thrombus Burden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other); Kaiping Central Hospital (Other); Second Affiliated Hospital of Shantou University Medical College (Other); The Third Xiangya Hospital of Central South University (Other); Sihui City People's Hospital (Unknown); Shenzhen Baoan District Shiyan People's Hospital (Unknown); People's Hospital of Nanxiong County (Unknown); Yuebei People's Hospital (Other); Weifang Medical University (Other); Wuzhou Gongren Hospital (Unknown); Dafeng Hospital of Chaoyang District in Shantou City (Unknown); Shenzhen Baoan People's Hospital (Unknown); Dongguan People's Hospital (Other Government); Yangchun People's Hospital (Unknown); Taishan People's Hospital (Unknown); The Second People's Hospital of Foshan (Other); Guangzhou Hospital of integrated Traditional and West Medicine (Unknown); Guangning People's Hospital (Unknown); Foshan Sanshui District People's Hospital (Unknown); Qingyuan People's Hospital (Other); Luhe County People's Hospital (Unknown); People's Hospital of Xinjiang Uygur Autonomous Region (Other); The Fourth People's Hospital of Chenzhou (Unknown); People's Hospital of Dapu County (Unknown); Shenzhen People's Hospital (Other); Heyuan people's Hospital (Unknown); Huaiji People's Hospital (Unknown); People's Hospital of Yingde City (Unknown); Qingyuan Hospital of Traditional Chinese Medicine Affiliated To Guangzhou University of Traditional Chinese Medicine (Unknown); Zhongshan Hospital Of Traditional Chinese Medicine (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); Lianzhou People's Hospital (Unknown); Lianping Xian Ren Ming Yi Yuan (Unknown); Guangxi Zhuang Autonomous Region Nationalities Hospital (Unknown); Liuzhou Municipal Liutie Central Hospital (Unknown); Chen Zhou 3RD People's Hospital (Unknown); Longgang District People's Hospital of Shenzhen (Other); The Affiliated Shunde Hospital of Jinan University (Unknown); Shenzhen Longhua District Central Hospital (Unknown); Shantou Central Hospital (Other); Tongxiang First People's Hospital (Unknown); Bobai County People's Hospital, Guangxi (Unknown); Meizhou Traditional Chinese Medicine Hospital (Unknown); The Third Affiliated Hospital of Sun Yat-Sen University, Yuedong Hospital (Unknown); Shenzhen Third People's Hospital (Other); Yangjiang People's Hospital (Other); Jiangmen Central Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); The First People's Hospital of Kashgar Erea (Unknown); First People's Hospital of Foshan (Other); Zhaoqing Gaoyao People's Hospital (Unknown); People's Hospital of Nanhai District, Foshan (Unknown); The Second Affiliated Hospital of Dalian Medical University (Other); Nanning Second People's Hospital (Other); The Second People's Hospital of Nanhai District of Foshan (Unknown); Shangyou People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDREC2018404H(R2)
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: Thrombus Aspiration; Coronary Intervention; Thrombus Burden; ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombus aspiration (Experimental): Upfront manual thrombus aspiration followed by PCI
  Interventions: Procedure: Thrombus aspiration
- PCI Alone (Active Comparator): PCI without upfront manual thrombus aspiration
  Interventions: Procedure: PCI Alone

INTERVENTIONS:
Procedure: Thrombus aspiration — Percutaneous Coronary Intervention with manual aspiration thrombectomy
  Arms: Thrombus aspiration
Procedure: PCI Alone — Percutaneous Coronary Intervention without manual aspiration thrombectomy
  Arms: PCI Alone

SUMMARY:
This is a prospective, multicenter, open-label, randomized, controlled, parallel group study, in which ST-segment Elevation Myocardial Infarction (STEMI) patients with high thrombus burden(TIMI thrombus grade ≥3) are included. Patients are randomized to be treated with or without manual thrombus aspiration(TA) during primary percutaneous coronary intervention(PPCI) by a ratio of 1:1.

DETAILED DESCRIPTION:
This study is intended to explore the efficacy of thrombus aspiration (TA) in ST-Segment Elevation Myocardial Infarction (STEMI) patients with high thrombus burden who received primary PCI within 12 hours after the onset of symptoms, reducing the incidence of cardiovascular death, recurrent myocardial infarction, stent thrombosis, target vessel revascularization within 180 days or stroke in 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. STEMI patients undergoing primary PCI within 12 hours after the onset of symptoms;
3. High thrombus burden after guidewire passes the lesion (TIMI thrombus grade ≥3);
4. Informed consent must be voluntary;

Exclusion Criteria:

1. Haemodynamic instability or cardiogenic shock;
2. After thrombolytic therapy;
3. The predicted survival time is less than 6 months due to non-cardiac disease;
4. History of coronary artery bypass grafting;
5. Participate in other researches within 30 days;
6. Preoperative gastrointestinal bleeding or contraindications to dual antiplatelet therapy;
7. Patients were considered unsuitable by other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3838 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | up to180 days
  The first occurrence of cardiovascular death, recurrent myocardial infarction, stent thrombosis or target vessel revascularization

SECONDARY OUTCOMES:
Stroke | up to 30 days
  The symptoms continuing for more than 24 hours or leading to death with no apparent cause other than vascular
Composite adverse cardiocerebrovascular events | up to 1 year
  The first occurence of cardiovascular death, recurrent myocardial infarction, stent thrombosis, target vessel revascularization or stroke.

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - First People's Hospital of Foshan, Foshan, Guangdong
  - The Second People's Hospital of Nanhai District, Foshan, Guangdong
  - First People's Hospital of Shunde (Affiliated Hospital at Shunde, Southern Medical University), Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - The first Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of traditional Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Huangpu Division of The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - Huizhou Third People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - The Second Affiliated Hospital of Shantou university Medical College, Shantou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Bao'an District People's Hospital, Shenzhen, Guangdong
  - Taishan people's Hospital, Taishan, Guangdong
  - Nanxiong people's Hospital, Xiongzhou, Guangdong
  - People's Hospital of Yangjiang City, Yangjiang, Guangdong
  - The Second Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Sihui people's Hospital, Zhaoqing, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital, Sun Yat-Sen University, Zhuhai, Guangdong
  - Zhuhai people's Hospital, Zhuhai, Guangdong
  - Guilin people's Hospital, Guilin, Guangxi
  - The Second Clinical College of Hainan Medical University, Haikou, Hainan
  - Hainan People's Hospital, Haikou, Hainan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - GanZhou Municopal Hospital, Ganzhou, Jiangxi
  - Shangyou Hospital, Ganzhou, Jiangxi
  - Affiliated Hospital, Weifang Medical University, Weifang, Shandong
  - The first Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Kashgar first people's Hospital, Kashgar, Xinjiang
  - The First Affilicated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - Shaoxing people's Hospital, Shaoxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrick JB. Landmark article (JAMA 1912). Clinical features of sudden obstruction of the coronary arteries. By James B. Herrick. JAMA. 1983 Oct 7;250(13):1757-65. No abstract available. PMID 6350634
- [Background] DeWood MA, Spores J, Notske R, Mouser LT, Burroughs R, Golden MS, Lang HT. Prevalence of total coronary occlusion during the early hours of transmural myocardial infarction. N Engl J Med. 1980 Oct 16;303(16):897-902. doi: 10.1056/NEJM198010163031601. PMID 7412821
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Beran G, Lang I, Schreiber W, Denk S, Stefenelli T, Syeda B, Maurer G, Glogar D, Siostrzonek P. Intracoronary thrombectomy with the X-sizer catheter system improves epicardial flow and accelerates ST-segment resolution in patients with acute coronary syndrome: a prospective, randomized, controlled study. Circulation. 2002 May 21;105(20):2355-60. doi: 10.1161/01.cir.0000016350.02669.1d. PMID 12021220
- [Background] Burzotta F, Trani C, Romagnoli E, Mazzari MA, Rebuzzi AG, De Vita M, Garramone B, Giannico F, Niccoli G, Biondi-Zoccai GG, Schiavoni G, Mongiardo R, Crea F. Manual thrombus-aspiration improves myocardial reperfusion: the randomized evaluation of the effect of mechanical reduction of distal embolization by thrombus-aspiration in primary and rescue angioplasty (REMEDIA) trial. J Am Coll Cardiol. 2005 Jul 19;46(2):371-6. doi: 10.1016/j.jacc.2005.04.057. PMID 16022970
- [Background] Vlaar PJ, Svilaas T, van der Horst IC, Diercks GF, Fokkema ML, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. Lancet. 2008 Jun 7;371(9628):1915-20. doi: 10.1016/S0140-6736(08)60833-8. PMID 18539223
- [Background] Frobert O, Lagerqvist B, Olivecrona GK, Omerovic E, Gudnason T, Maeng M, Aasa M, Angeras O, Calais F, Danielewicz M, Erlinge D, Hellsten L, Jensen U, Johansson AC, Karegren A, Nilsson J, Robertson L, Sandhall L, Sjogren I, Ostlund O, Harnek J, James SK; TASTE Trial. Thrombus aspiration during ST-segment elevation myocardial infarction. N Engl J Med. 2013 Oct 24;369(17):1587-97. doi: 10.1056/NEJMoa1308789. Epub 2013 Aug 31. PMID 23991656
- [Background] Jolly SS, Cairns JA, Yusuf S, Meeks B, Pogue J, Rokoss MJ, Kedev S, Thabane L, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Steg PG, Bernat I, Xu Y, Cantor WJ, Overgaard CB, Naber CK, Cheema AN, Welsh RC, Bertrand OF, Avezum A, Bhindi R, Pancholy S, Rao SV, Natarajan MK, ten Berg JM, Shestakovska O, Gao P, Widimsky P, Dzavik V; TOTAL Investigators. Randomized trial of primary PCI with or without routine manual thrombectomy. N Engl J Med. 2015 Apr 9;372(15):1389-98. doi: 10.1056/NEJMoa1415098. Epub 2015 Mar 16. PMID 25853743
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Background] Jolly SS, James S, Dzavik V, Cairns JA, Mahmoud KD, Zijlstra F, Yusuf S, Olivecrona GK, Renlund H, Gao P, Lagerqvist B, Alazzoni A, Kedev S, Stankovic G, Meeks B, Frobert O. Thrombus Aspiration in ST-Segment-Elevation Myocardial Infarction: An Individual Patient Meta-Analysis: Thrombectomy Trialists Collaboration. Circulation. 2017 Jan 10;135(2):143-152. doi: 10.1161/CIRCULATIONAHA.116.025371. Epub 2016 Dec 9. PMID 27941066
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621